CLINICAL TRIAL: NCT06636656
Title: Phase IIa, Single-arm, Open-label, Multi-center Clinical Trial to Evaluate the Efficacy, Safety, and Tolerability of Intravenous Induction and Subcutaneous Maintenance Treatment With BI 3032950 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: A Study to Test Whether BI 3032950 Helps People With Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1486-0006; 2023-509544-10-00 (Registry Identifier: CTIS (EU)); U1111-1300-3640 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: The study consists of Part A and Part B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will receive an intravenous dose of BI 3032950 in Part A followed by a subcutaneous dose of BI 3032950 in Part B.
  Interventions: Drug: BI 3032950 intravenous (Part A); Drug: BI 3032950 subcutaneous (Part B)

INTERVENTIONS:
Drug: BI 3032950 intravenous (Part A) — BI 3032950 intravenous (Part A)
Drug: BI 3032950 subcutaneous (Part B) — BI 3032950 subcutaneous (Part B)

SUMMARY:
Adults between 18 and 80 years of age with ulcerative colitis can participate in this study. This is a study for people for whom previous treatment was not successful or who stopped previous treatment. The purpose of this study is to find out whether BI 3032950 helps people with ulcerative colitis.

This study has 2 parts. In Part A, participants get BI 3032950 as an infusion into a vein every 4 weeks. After 12 weeks, doctors check whether the signs and symptoms of ulcerative colitis have improved. Before the results of this assessment are available, participants move on to Part B and get BI 3032950 as an injection under the skin. Participants whose results show clinical response after 12 weeks can continue treatment with BI 3032950. They get BI 3032950 injections under the skin every 4 weeks for up to 2 years.

Participants visit their doctors every 4 weeks. During these visits, the doctors check the signs and symptoms of ulcerative colitis. This includes taking blood and stool samples. Doctors also do endoscopies. This is a procedure that uses a tube with a camera to look inside the body.

The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Female and male participants aged 18 to 80 years (inclusive) at the time of informed consent,
* Diagnosis of ulcerative colitis (UC) ≥3 months prior to screening by clinical and endoscopic evidence corroborated by a histopathology report,
* Inadequate response, loss of response, or intolerance to treatment with biologic/targeted therapy or termination of treatment with biologic/targeted therapy for any other reason,
* Female participants of childbearing potential must be ready and able to use highly effective methods of birth control and male participants are required to use condoms,
* Further inclusion criteria apply.

Exclusion criteria

* Diagnosis of indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, microscopic colitis, or Crohn's disease (CD),
* Findings suggestive of CD (e.g. fistulae, granulomas on biopsy),
* Evidence of colonic moderate/severe mucosal dysplasia or colonic adenomas, unless properly removed,
* Gastrointestinal neoplasia, primary sclerosing cholangitis, or known colonic stricture,
* Evidence of fulminant colitis or toxic megacolon at screening,
* Current ileal-pouch anal anastomosis, ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine,
* Previous surgery or anticipated surgical intervention for UC (trial participants with previous colonic surgery may be allowed based on investigator's judgement after discussion with the sponsor),
* Any current or prior abscesses, unless they have been drained and treated at least 6 weeks prior to first trial drug administration and are not anticipated to require surgery,
* Further exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with clinical remission defined by the modified Mayo Score [mSC] with mSC of 0 to 2, including stool frequency subscore [SFS] of 0 or 1, rectal bleeding subscore [RBS] of 0, and centrally-read endoscopy subscore [ESS] of 0 or 1 | Up to Week 12
  The modified Mayo score (mMS) consists of 3 components
  1. Stool frequency subscore (SFS)
  2. Rectal bleeding subscore (RBS)
  3. Endoscopy subscore (ESS) Each component is graded from 0 = none to 3 = severe. The overall range of the mMS is from 0 to 9 with a higher score indicating a worsening of the symptoms.

SECONDARY OUTCOMES:
Endoscopic remission (defined as centrally-read ESS of 0) | Up to Week 12
  The endoscopy subscore (ESS) is graded from 0 = none to 3 = severe. The ESS is part of the modified Mayo score.
Clinical response (defined as a decrease from baseline in mMS ≥2 and at least a 30% reduction from baseline, and a decrease in RBS of ≥1 or an absolute RBS of 0 or 1) | Up to Week 12
  The modified Mayo score (mMS) consists of 3 components
  1. Stool frequency subscore (SFS)
  2. Rectal bleeding subscore (RBS)
  3. Endoscopy subscore (ESS) Each component is graded from 0 = none to 3 = severe. The overall range of the mMS is from 0 to 9 with a higher score indicating a worsening of the symptoms.
Endoscopic improvement (defined as centrally-read ESS of 0 or 1) | Up to Week 12
  The endoscopy subscore (ESS) is graded from 0 = none to 3 = severe. The ESS is part of the modified Mayo score.
Modified Mayo Score change from baseline | Up to Week 12
  The modified Mayo score (mMS) consists of 3 components
  1. Stool frequency subscore (SFS)
  2. Rectal bleeding subscore (RBS)
  3. Endoscopy subscore (ESS) Each component is graded from 0 = none to 3 = severe. The overall range of the mMS is from 0 to 9 with a higher score indicating a worsening of the symptoms.
Stool frequency subscore of 0 or 1 | Up to Week 12
  The stool frequency (SFS) is graded from 0 = none to 3 = severe. The SFS is part of the modified Mayo score.
Rectal bleeding subscore of 0 | Up to Week 12
  The rectal bleeding subscore (RBS) is graded from 0 = none to 3 = severe. The RBS is part of the modified Mayo score.
Occurrence of treatment-emergent adverse events (AEs) | Up to Week 12 and up to Week 104

CONTACTS AND LOCATIONS:
Locations (42):
- United States (14):
  - One of a Kind Clinical Research Center, Scottsdale, Arizona
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Clinical Research of Osceola, Kissimmee, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Illinois Gastroenterology Group - Gurnee, Gurnee, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Columbia University Medical Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Texas Digestive Disease Consultants, Cedar Park, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington
  - Digestive Health Specialists, Tacoma, Washington
- Belgium (2):
  - UZ Leuven, Leuven
  - CHC MontLegia, Liège
- Czechia (2):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - ISCARE a.s., Prague
- Poland (15):
  - Centrum Medyczne Plejady, Krakow
  - Medrise Sp. z o.o., Lublin
  - Eskulap Pabianice Sp. z o.o., Pabianice
  - EMC Instytut Medyczny S.A. - Poznan 70-304, Poznan
  - Clinical Research Center Sp. z o.o. Medic-R sp.k., Poznan
  - Centrum Medyczne Medyk Sp. z o.o., Rzeszów
  - Endoskopia Sp. z o.o., Sopot
  - Twoja Przychodnia Szczecinskie Centrum Medyczne Sp. z o.o., Szczecin
  - Gastromed Sp. z o.o., Torun
  - Synexus Polska Sp. z o.o., Warsaw
  - NZOZ VIVAMED Jadwiga Miecz, Warsaw
  - PlanetMed Sp. z o.o., Wroclaw
  - EMC Instytut Medyczny S.A. - Wroclaw, Wroclaw
  - Centrum Diagnostyczno Lecznicze Barska Sp. z o.o., Włocławek
  - Pro Life Medica Sp. z o.o., Zamość
- Serbia (4):
  - Clinical Hospital Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Zemun, Belgrade
  - General Hospital - Djordje Joanovic, Zrenjanin
- Slovakia (5):
  - F D Roosevelt University General Hospital Of Banska Bystrica, Banská Bystrica
  - ENDOMED s.r.o., Košice
  - KM Management, spol. s.r.o., Nitra
  - Gastro I., s.r.o, Prešov
  - Accout Center s.r.o., Šahy

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com